CLINICAL TRIAL: NCT02341261
Title: Activity for Diabetic Polyneuropathy: the ADAPT Study
Brief Title: Activity for Diabetic Polyneuropathy
Acronym: ADAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of Kansas (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20015791; R01DK064814 (NIH)
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care Counseling (Experimental): Participants randomized to the control group will receive diet and exercise counseling at baseline and 9 months. Participants will wear an ActivePAL for 7 days at baseline, 9 months, and 18 months without stimulation.
  Interventions: Behavioral: Standard Care Counseling
- Supervised Exercise and Counseling (Experimental): Participants randomized to the intervention will perform supervised aerobic, resistance and balance training twice weekly for 12 weeks, and weekly thereafter. Actigraphy-based counseling to reduce sedentary behavior will follow a similar taper. Daily text messages, "tweets", emails, and social media posts at random times during waking hours will be used to provide reminders and motivational messages. Participants will have 11 separate 7-day continuous ActivePAL training session incorporating vibrostimulatory feedback spread across the treatment period.
  Interventions: Behavioral: Supervised Exercise and Counseling

INTERVENTIONS:
Behavioral: Standard Care Counseling
  Arms: Standard Care Counseling
Behavioral: Supervised Exercise and Counseling
  Arms: Supervised Exercise and Counseling

SUMMARY:
The proposed study will randomize participants with diabetic peripheral neuropathy into two groups. One group of participants will receive standard-of-care counseling while the other group will undergo supervised exercise and counseling to increase physical activity.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) affects over 8% of Americans, and half will develop peripheral neuropathy, a progressive injury to the very longest nerves of the body. Our previous research has found that neuropathy can be detected early in its course and followed by examining nerves that reach to the skin using a small punch biopsy. These cutaneous nerves can be injured by high blood glucose, obesity and high triglycerides, but have the potential to regrow in response to treatments that improve these metabolic conditions. The proposed study will randomize participants with mild to moderate diabetic peripheral neuropathy to receive either generic annual counseling or an integrated program of moderate supervised exercise and actigraphy based anti sedentariness counseling.

ELIGIBILITY:
Inclusion Criteria:

1. T2D defined by ADA criteria.
2. Peripheral neuropathy based on the Toronto Diabetic Neuropathy Expert Group consensus criteria for "Confirmed diabetic sensorimotor peripheral neuropathy".
3. Moderate DPN severity with a UENS of 2-18.
4. Age between 30 and 75.
5. Under the care of an identified Primary Care Physician (PCP).

Exclusion Criteria:

1. Any alternative cause for peripheral neuropathy. The following tests must have been found normal within the last 12 months or will be performed pre-randomization: vitamin B12, serum protein electrophoresis and immunofixation. ANA and TSH may be obtained if clinically indicated and not available from clinical records.
2. Family history of a non-diabetic neuropathy in a first-degree relative.
3. Severe or longstanding neuropathy: UENS > 18 or history of foot ulceration or amputation.
4. Participants taking Coumadin or oral factor X or thrombin inhibitor therapy will be considered on an individual basis by the site investigator.
5. Severe edema, dermatologic or lower extremity condition that would increase risk of skin biopsy.
6. A serious medical condition that might shorten life span or prevent exercise.
7. Subjects with obesity or hypertension considered in a dangerous range (BMI> 45, systolic BP >170, or diastolic BP >110) and those who fail a medically supervised graded maximal stress test will be excluded from the study for safety reasons.
8. An inability to understand or cooperate with the procedures of the study
9. Females who are pregnant at screening or actively plan to become pregnant during the study period, because of the marked changes in metabolism anticipated during pregnancy.
10. If ,in the investigators assessment, that participation in the study would be limited by a person's weight, size, or other physical condition.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-11; Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change in Intraepidermal Nerve Fiber Density (IENFD) | Baseline, 9 months, and 18 months
Change in Quality of Life (NQOL-DN) Questionnaire Results | Baseline, 9 months, and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: A. Gordon Smith, MD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - University of Kansas, Kansas City, Kansas
  - University of Utah School of Medicine, Salt Lake City, Utah

REFERENCES:
- [Derived] Kluding PM, Singleton JR, Pasnoor M, Dimachkie MM, Barohn RJ, Smith AG, Marcus RL. Activity for Diabetic Polyneuropathy (ADAPT): Study Design and Protocol for a 2-Site Randomized Controlled Trial. Phys Ther. 2017 Jan 1;97(1):20-31. doi: 10.2522/ptj.20160200. PMID 27417167